CLINICAL TRIAL: NCT06182592
Title: A Randomized, Multi-center, Open-label Phase III Bridging Study to Compare Efficacy of Liposomal Cytarabine-Daunorubicin for Injection With Cytarabine and Daunorubicin in Treating Older Patients With High-Risk (Secondary) Acute Myeloid Leukemia
Brief Title: A Bridging Study of Liposomal Cytarabine-Daunorubicin in Treating Olderly Patients With Treatment-naive High-Risk (Secondary) Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC1702-004
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: High-risk (Secondary) Acute Myeloid Leukemia
MeSH Terms: conditions — Neoplasm Metastasis; Leukemia, Myeloid, Acute | interventions — Injections; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (liposomal cytarabine-daunorubicin for injection) (Experimental): Patients are eligible to receive up to 2 inductions and up to 2 consolidations with liposomal cytarabine-daunorubicin for injection. The number of inductions and consolidations a patient received will depend on response.
  Interventions: Drug: Liposomal cytarabine-daunorubicin for injection
- Arm B (7+3) (Experimental): Patients are eligible to receive up to 2 inductions and up to 2 consolidations with cytarabine and daunorubicin given as a 7+3, or 5 days of continuous infusion of cytarabine and 2 days of daunorubicin (5+2, second induction, consolidation courses) therapy. The number of inductions and consolidations a subject received will depend on response.
  Interventions: Drug: 7+3 (cytarabine and daunorubicin)

INTERVENTIONS:
Drug: Liposomal cytarabine-daunorubicin for injection — First induction: 100 units/m^2 by 90-minute IV infusion on Days 1, 3, 5. Second induction: 100 units/m^2 by 90-minute IV infusion on Days 1 and 3. Consolidation therapy: 65 units/m^2 by 90-minute IV infusion on Days 1 and 3.
  Arms: Arm A (liposomal cytarabine-daunorubicin for injection)
Drug: 7+3 (cytarabine and daunorubicin) — First induction: 7+3 will be administered as: cytarabine at a dose of 100 mg/m^2/day on Days 1 through 7 by continuous infusion, and daunorubicin at a dose of 60 mg/m^2/day on Days 1, 2, and 3.
  Second induction: 5+2 will be administered as: cytarabine at a dose of 100 mg/m^2/day on Days 1 through 5 by continuous infusion and daunorubicin at a dose of 60 mg/m^2/day on Days 1 and 2.
  Consolidation therapy: 5+2 will be administered as: cytarabine at a dose of 100 mg/m^2/day on Days 1 through 5 by continuous infusion, and daunorubicin at a dose of 60 mg/m^2/day on Days 1 and 2.
  Arms: Arm B (7+3)

SUMMARY:
The purpose of this bridging study is to determine the efficacy of liposomal cytarabine-daunorubicin for injection compared with cytarabine and daunorubicin in older patients with high-risk (secondary) acute myeloid leukemia.

DETAILED DESCRIPTION:
Liposomal cytarabine-daunorubicin for injection manufactured by CSPC Zhongnuo Pharmaceutical Technology Co., Ltd is a class 3 chemical drug imitating Vyxeos developed by Jazz Pharmaceuticals plc. This bridging trial compares the efficacy of liposomal cytarabine-daunorubicin for injection manufactured by CSPC Zhongnuo Pharmaceutical Technology Co., Ltd with cytarabine/daunorubicin (7+3) in elderly patients with treatment-naïve high-risk (secondary) AML to determine that test drug is comparable to Vyxeos in efficacy, safety and pharmacokinetic properties. Patients will be randomized in a 1:1 ratio to receive liposomal cytarabine-daunorubicin or daunorubicin/cytarabine as induction and consolidation chemotherapy. Patients will receive up to two cycles of induction and consolidation therapy. After the treatment period, there is a follow-up phase for overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and voluntarily sign informed consent.
* Male or female between 60-75 years of age (inclusive).
* Pathological diagnosis of AML according to 2022 WHO criteria (with at least 20% blasts in the peripheral blood or bone marrow) and fulfill of one of the following standards:

  1. Therapy related AML: t-AML must have a documented history of prior cytotoxic therapy or ionizing radiotherapy for an unrelated disease;
  2. AML with a history of myelodysplasia: MDSAML must have bone marrow documentation of prior MDS;
  3. AML with a history of CMMoL: CMMoLAML must have bone marrow documentation of prior CMMoL;
  4. De novo AML with karyotypic abnormalities characteristic of MDS: de novoAML must have cytogenetics with abnormalities per WHO.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Laboratory values meet the following criteria:

  1. Serum creatinine≤2 × ULN;
  2. Serum total bilirubin≤2 × ULN, ≤3 × ULN for patients with liver involvement;
  3. Serum alanine aminotransferase or aspartate aminotransferase≤3 × ULN, ≤5 × ULN for patients with liver involvement.
* Cardiac function (LVEF) ≥ 50% by echocardiography or MUGA.
* QTcF (Fridericia's) for male<450 ms, for female<470 ms at screening.
* Male and female of childbearing potential must agree to use contraceptive measures (such as IUD, contraceptive or condom) during the study and within 6 months after the end of the study.

Exclusion Criteria:

* Acute promyelocytic leukemia; or favorable cytogenetics, including t(8;21) or inv16 if known at the time of randomization.
* Except for CMMoL, patients with history of myeloproliferative neoplasms (MPN) (defined as a history of essential thrombocytosis or polycythemia vera, or idiopathic myelofibrosis prior to the diagnosis of AML) or combined MDS/MPN are not eligible.
* History of other malignancy within 3 years before randomization, expect for cancers that have been cured (basal cell or squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of cervix and breast or prostate cancer with Gleason score of 6).
* Patients with clinical evidence of active CNS leukemia.
* Prior treatment for AML (except for hydroxyurea) or stem-cell transplantation.
* Administration of any therapy for MDS (conventional or investigational) within 2 weeks prior to of the first dose of study drug; use of hydroxyurea for the purpose of inhibiting rapid tumor proliferation within 24 hours before the first dose. Toxicities associated with prior MDS therapy have not recovered to grade 1 or less prior to start of treatment.
* Any major surgery or radiation therapy within 4 weeks.
* Patients with previous cumulative exposure to anthracyclines >368 mg/m^2 daunorubicin (or equivalent drug equivalent dose level).
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent.
* Patients with myocardial impairment of any cause (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by NYHA Criteria (Class Ш or Ⅳ staging).
* Active or uncontrolled infection.
* Current evidence of invasive fungal infection (blood or tissue culture).
* Patients with known HIV, hepatitis B or hepatitis C infection.
* Patients who are hypersensitive to cytarabine, daunorubicin or liposomal products.
* Patients with a history of Wilson's disease or other copper-metabolism disorders.
* Participation in another clinical trial or treatment with any investigational drug within 28 days prior to screening.
* Any patients whom the investigator believes will not be a good candidate for the study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  Overall survival will be measured from the date of randomization to death from any cause.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 2 years
  EFS is defined as the time from study randomization to the date of induction treatment failure (persistent disease), relapse from complete remission (CR) or complete remission with incomplete count recovery (CRi) or death from any cause, whichever occurs first.
Duration of remission (DoR) | Up to 2 years
  DoR is defined as the time from the day achieving CR or CRi to the date of relapse or death. Only patients achieving CR or CRi will be assessed for remission duration.
CR rate | Up to 2 years
  Proportion of patients with complete remission during the treatment period.
Composite remission rate | Up to 2 years
  Proportion of patients with CR or CRi.
Proportion of patients receiving a haematopoietic stem cell transplant (HSCT) | Up to 2 years
  The number and percentage of patient transferred for HSCT after induction treatment will be recorded.
Proportion of pateints who achieve CR with MRD negativity | Up to 2 years
  The number and percentage of patients who are MRD negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Hospital of Blood Disease, Chinese Academy of Medical Sciences, Tianjin, China